CLINICAL TRIAL: NCT01949831
Title: The Effect of Systematic Assessment of Functional Ability, Development of Rehabilitation Plan and Follow-up at Home for Elderly Medical Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to inclusion problems (not recruting enough participants) recruiting participants has halted prematurely and will not resume.
Sponsor: Aarhus University Hospital (Other)
Collaborators: VIA University College (Other); Institute of public health, department of nursing sciences, Århus University, Denmark (Other)
Responsible Party: Principal Investigator, Louise Møldrup Nielsen, PhD student, occupational therapist, Aarhus University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MVAprojekt
Record Dates: First submitted 2013-09-13; First posted 2013-09-25 (Estimated); Last update posted 2014-03-03 (Estimated); Status verified 2014-02

CONDITIONS: Geriatric Disorder
Keywords: functional assessment; acute care; older medical patients

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Usual care
- Functional assessment (Experimental): Assessment of functional ability in combination with follow-up at home
  Interventions: Other: Assessment of functional ability in combination with follow-up at home

INTERVENTIONS:
Other: Assessment of functional ability in combination with follow-up at home
  Arms: Functional assessment

SUMMARY:
The aim of this study is to examine the effect of systematic assessment of functional ability, development of rehabilitation plan and follow-up at home for elderly medical patient's risk of readmission. The effect of the intervention is examined in a randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to, Medical Visitation Section (MVA) Aarhus University Hospital
* aged 65+
* resident in City of Aarhus.

Exclusion Criteria:

* Patients admitted from a psychiatric institution or nursing home
* patients without walking ability
* patients who do not speak or read Danish
* terminally ill patients
* patients transferred to other hospital departments

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 52 (Actual)
Dates: Start 2013-10; Primary Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Re-admission | Re-admission in 26 weeks
  *Primary outcome was originally set to readmissions within 26 weeks but due to clerical error it has been written as 30 days. The error has now been corrected.

SECONDARY OUTCOMES:
Mortality | 30 day mortality
Functional ability | 4 and 26 weeks after intervention
  Functional ability measured with World Health Organization Disability Assessment Schedule (WHODAS 2.0) and Barthel-20
Re-admission | Re-admission within 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Hans Kirkegaard, Professor, Principal Investigator — Center for Acute research
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark